CLINICAL TRIAL: NCT02509312
Title: A Prospective, Randomized, Control Trial of Ketorolac Versus Placebo on Opioid Analgesic Use, Estimated Blood Loss and Complications Following Cesarean Delivery With Epidural Morphine
Brief Title: Prospective Effect of Intravenous Ketorolac on Opioid Use, EBL and Complications Following Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, John J. Kowalczyk, Instructor of Anaesthesia - Beth Israel Deaconess Medical Center, Harvard Medical School / Harvard Medical School, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ketorolac-1
Record Dates: First submitted 2015-06-11; First posted 2015-07-28 (Estimated); Results first posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-05

CONDITIONS: Analgesia, Obstetrical; Postpartum Hemorrhage; Opioid Use; Nonsteroidals (NSAIDs)Toxicity; Coagulation Defect; Postpartum; Postoperative Pain; Ketorolac Adverse Reaction; Blood Loss, Postoperative
Keywords: Analgesia, Obstetrical; Blood Loss, Surgical; Analgesics, Opioid/administration & dosage; Cyclooxygenase Inhibitors/administration & dosage; Cesarean Delivery; Female; Humans; Ketorolac/administration & dosage; Hydromorphone/administration & dosage; Pain, Postoperative/drug therapy; Pregnancy; Morphine/administration & dosage; Cesarean Section Complications; Ketorolac
MeSH Terms: conditions — Agnosia; Postpartum Hemorrhage; Hemostatic Disorders; Pain, Postoperative; Postoperative Hemorrhage; Blood Loss, Surgical; Pain | interventions — Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo (normal saline) or ketorolac in syringe prepared by the investigational pharmacy with study kit number and blinding key maintained by investigational pharmacy until time of unblinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental (Experimental): Patients in this arm will be given ketorolac at cord clamp with standard dose of 30 mg, then 3 additional 30 mg doses every 6 hours
  Interventions: Drug: Ketorolac
- Control (Placebo Comparator): Patients in this arm will be given a placebo medication at cord clamp, and then 3 additional doses of placebo every 6 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketorolac — Patients in the experimental arm will receive ketorolac 30 mg in 1 ml at the time of cord clamp and then for 3 more doses every 6 hours.
  Other Names: Toradol
  Arms: Experimental
Drug: Placebo — Patients in the control arm will receive normal saline 1 ml at the time of cord clamp and then for 3 more doses every 6 hours.
  Arms: Control

SUMMARY:
In this randomized, double-blind control trial to evaluate the effect of ketorolac given at the time of cord clamp has on estimated blood loss and postcesarean pain control. Patients will be randomized to either placebo or ketorolac prior to surgery. Those randomized to ketorolac will receive ketorolac at cord clamp and three additional doses every 6 hours (total 4 doses/24 hours). Those in the placebo group will receive normal saline during those time periods. Our primary outcome is to assess whether intra-operative ketorolac increases the estimated blood loss during Cesarean delivery.

DETAILED DESCRIPTION:
Background:

Opioid analgesics are among the most common medication employed for post-cesarean delivery pain management. However, opioid side-effects such as, nausea, vomiting, urinary retention, and sedation are problematic and can adversely impact post-operative recovery. Non-steroidal anti-inflammatory medications have analgesic as well as anti-inflammatory properties making them an ideal alternative for opioid analgesics. Ketorolac, which can be given by either oral and parenteral routes, is frequently employed as a post-surgical analgesic in a variety of procedures including gynecologic and obstetric, and has comparable analgesic properties to opioids without the aforementioned side-effects.(1)

Additionally, two studies have specifically evaluated administration of ketorolac in the treatment of post-cesarean section pain in patients receiving either patient controlled intravenous analgesia or patient controlled epidural analgesia.(2, 3) However, due to the known inhibition of prostaglandin synthesis, several retrospective and observational studies have suggested that ketorolac and other non-steroidal anti-inflammatory drugs (NSAIDs) may be associated with an increase in estimated blood loss (EBL) and uterine atony.(4,5) This research showed in vivo defects in platelet function, however a recent meta-analysis in a variety of different surgical procedures suggest there is no clinically significant difference in EBL attributed to the administration of ketorolac compared to placebo.(6)

Despite this, there still exists significant resistance to the intraoperative and post-operative use of ketorolac due to concerns of increasing EBL. This is particularly true with regard to cesarean sections, which, due to the nature of the procedure is associated with an EBL higher than found in many other surgeries and possibly leading to increased morbidity. To our knowledge there have only been three previous studies that specifically examined the use of ketorolac with cesarean delivery.

El-Tahan et al, administered ketorolac preoperatively and focused on the blunting of sympathetic response to intubation of healthy patients undergoing cesarean section under general anesthesia. This study evaluated only a single low dose followed by intraoperative infusion. Although they did look at intraoperative EBL, they did not give additional postoperative doses or assess postoperative bleeding.(7) Lowder et al and Pavy et al looked at postoperative use of ketorolac on pain control and EBL, but no intraoperative dose of ketorolac was given.(2,3)

To our knowledge, there have been no studies that evaluated intraoperative ketorolac on post-operative opioid analgesic use and EBL during cesarean delivery with epidural analgesia and intra-epidural administration of morphine.

Screening/Eligibility Visit:

Patients admitted to MacDonald Women's Hospital for scheduled or non-scheduled, non-urgent Cesarean delivery will be screened for potential eligibility. Potential participants will be then be approached to confirm they meet inclusion and exclusion requirements. Patients will then be consented with an IRB-approved informed consent prior to enrollment.

Randomization & Blinding:

Patients will be randomized to receive either ketorolac 30 mg in 1 ml (n=35) or normal saline 1 ml (n=35). Randomization will be performed by the Investigational Pharmacy in a block of four design. No one involved with patient care, enrollment or data collection will have access to the unblinding key until completion of the study. The randomization key will be kept in the Investigational Research Pharmacy, and they will prepare the medications accordingly. Upon arrival in the OR, the anesthesiologist will open an envelope that will contain the kit number corresponding to the patient's study identification number. The anesthesiologist or anesthetist will remove the assigned kit from the Omnicell. Patients, clinicians and study staff will be unaware of the patient's assigned study group. Upon study completion by all patients, the randomization key will be provided to the study staff upon request.

Brief Study Methods:

After obtaining written informed consent, the Investigation Research Pharmacy an envelope that will contain the kit number corresponding to the patient's study identification number. Basic demographic information is collected from the patient. Each patient will undergo combined spinal-epidural anesthesia with our standard cesarean induction dose of hyperbaric 0.75% bupivacaine 1.5 ml intrathecally and fentanyl 100mcg epidurally. The patient will be moved to the supine position with left lateral uterine displacement. When a T6 sensory level to pinprick is achieved, Cesarean delivery will proceed using the standard procedures established in our institution. Once the newborn is delivered and the cord is clamped, the first dose of the ketorolac/placebo will be administered by the anesthesiologist or anesthetist. Any additional medications required for sedation or pain control during the remainder of the surgery (hydromorphone and acetaminophen) will be given, as appropriate for patient comfort. Prior to the completion of the procedure, the patient will receive epidural morphine 3 mg per the standard protocols. Postoperatively, the patient will receive the corresponding three additional scheduled doses of ketorolac/placebo every 6 hours. Supplemental analgesia will be administered according to a standard post-operative pain management protocol on labor and delivery with acetaminophen and intravenous hydromorphone provided, as needed for pain control.

Exposures and their measurement:

Exposure: Ketorolac 30 mg IV or Normal Saline 1 ml (Placebo) IV

Measurements: See outcomes and their measurements

Outcomes and their measurement:

Primary outcome: Estimated Blood Loss (EBL) will be compared between groups. Secondary outcomes: Rate of Post-Partum Hemorrhage, Corrected Change in Hct on POD1, Uterotonic Doses, Units of Packed Reb Blood Cell Transfused, Hydromorphone Use, Total Hydromorphone Dose, Anti-emetic Doses, Pruritus Doses, Percentile Change in Systolic Blood Pressure at 6, 12, and 24 hours, Percentile Change in Diastolic Blood Pressure at 6, 12, and 24 hours, and Pain score at 0 and 15 minutes and 1, 6, 12 and 24 Hours post-Cesarean Delivery.

Confounders and their measurement:

Many confounders should be limited by the nature of an RCT in a select patient population and pre- and intra-operative exclusion criteria. Additional potential confounders, including intraoperative fluid volume administration and patient adherence to study medication, will be recorded. Posthoc analysis will be performed to determine if any differences between groups were significant.

Analysis plan:

Data will be assessed for normality using histograms, QQ plots and Shapiro-Wilk test. Demographic, obstetric, and perioperative data will be presented as mean (standard deviation), median [interquartile range] or count (percentage), as appropriate. Between-group comparisons will be assessed using the t-test and Wilcoxon signed-rank test, as appropriate. For dichotomized outcomes, a Chi-square test will be performed to assess the proportions between groups.

Sample size justification:

A priori power analysis was performed to determine the sample size. Based on our prior retrospective study, we knew that the mean estimated blood loss for uncomplicated Cesarean deliveries was 814 ml with a standard deviation of 242 ml. We set our difference between groups to 186 ml. This would detect an EBL of >1,000 ml in the ketorolac group, a value large enough to classify the ketorolac group as post-partum hemorrhage and potentially escalate care and lead to additional maternal morbidity. With an alpha error of 0.05 and a power of 80%, we estimated that a sample size of 28 patients per group would be needed or 56 total patients enrolled. We had concern for loss after enrollment due to acuity, cases after 4 pm and exclusion criteria including intraoperative EBL and obstetric refusal. We planned for the loss of 20% of enrolled patients and increased the total study enrollment number to 70.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a scheduled or non-scheduled, non-urgent primary or repeat Cesarean delivery between 37-42 weeks gestational age,
* Viable singleton intra-uterine pregnancy,
* Patients undergoing a scheduled or unscheduled, non-emergent/non-urgent Cesarean delivery for placenta previa or vasa previa,
* Neuraxial anesthesia with combined spinal-epidural placed for surgery,
* Patients must be 18 years or older as well as willing and able to provide informed consent.

Exclusion Criteria:

* Patients unable or unwilling to provide informed consent,
* Urgent or emergent Cesarean delivery
* Multiple fetal gestations (>1 intrauterine pregnancy),
* Cesarean delivery for bleeding such as placental abruption or actively bleeding placenta previa or vasa previa,
* Contraindication to NSAID use eg: allergy, chronic renal disease,
* Patients with acute or chronic platelet dysfunction (e.g.: idiopathic thrombocytopenic purpura, HELLP syndrome),
* Platelets <100k,
* History of peptic ulcer disease,
* Inherited or acquired coagulopathies or bleeding disorder, (disseminated intravascular coagulopathy, hemophilia),
* Suspected or proven placenta accreta, increta or percreta,
* Inability to receive epidural morphine,
* Diagnosed chronic pain disorder on chronic adjunct or opioid analgesia,
* Use of general anesthesia during procedure.

Intraoperative exclusion criteria:

- EBL > 1000 ml prior to cord clamp

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blackburn A, Stevens JD, Wheatley RG, Madej TH, Hunter D. Balanced analgesia with intravenous ketorolac and patient-controlled morphine following lower abdominal surgery. J Clin Anesth. 1995 Mar;7(2):103-8. doi: 10.1016/0952-8180(94)00040-b. PMID 7598916
- [Background] Diemunsch P, Alt M, Diemunsch AM, Treisser A. Post cesarean analgesia with ketorolac tromethamine and uterine atonia. Eur J Obstet Gynecol Reprod Biol. 1997 Apr;72(2):205-6. doi: 10.1016/s0301-2115(96)02682-6. No abstract available. PMID 9134403
- [Background] Pavy TJ, Paech MJ, Evans SF. The effect of intravenous ketorolac on opioid requirement and pain after cesarean delivery. Anesth Analg. 2001 Apr;92(4):1010-4. doi: 10.1097/00000539-200104000-00038. PMID 11273941
- [Background] Lowder JL, Shackelford DP, Holbert D, Beste TM. A randomized, controlled trial to compare ketorolac tromethamine versus placebo after cesarean section to reduce pain and narcotic usage. Am J Obstet Gynecol. 2003 Dec;189(6):1559-62; discussion 1562. doi: 10.1016/j.ajog.2003.08.014. PMID 14710063
- [Background] El-Tahan MR, Warda OM, Yasseen AM, Attallah MM, Matter MK. A randomized study of the effects of preoperative ketorolac on general anaesthesia for caesarean section. Int J Obstet Anesth. 2007 Jul;16(3):214-20. doi: 10.1016/j.ijoa.2007.01.012. Epub 2007 Apr 24. PMID 17459695
- [Background] Elhakim M, Fathy A, Amine H, Saeed A, Mekawy M. Effect of i.v. tenoxicam during caesarean delivery on platelet activity. Acta Anaesthesiol Scand. 2000 May;44(5):555-9. doi: 10.1034/j.1399-6576.2000.00512.x. PMID 10786742
- [Background] Gobble RM, Hoang HLT, Kachniarz B, Orgill DP. Ketorolac does not increase perioperative bleeding: a meta-analysis of randomized controlled trials. Plast Reconstr Surg. 2014 Mar;133(3):741-755. doi: 10.1097/01.prs.0000438459.60474.b5. PMID 24572864

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketorolac: Patients in this arm will be given ketorolac at cord clamp with standard dose of 30 mg, then 3 additional 30 mg doses every 6 hours.
  Ketorolac: Patients in experimental arm will receive ketorolac 30 mg in 1 ml at time of cord clamp and then for 3 more doses every 6 hours.
  Epidural Morphine: All patients, including those in both the experimental and control groups, in this study will receive epidural morphine prior to removal of epidural catheter as part of routine obstetric care for cesarean delivery.
  Hydromorphone: Post-operatively all patients patients will have intravenous hydromorphone on an as needed basis to control their pain, as part of routine obstetric care for cesarean delivery.
- Placebo: Patients in this arm will be given a placebo medication at cord clamp, and then 3 additional doses of placebo every 6 hours.
  Placebo: Patients in the control arm will receive 1 ml of normal saline at time of cord clamp and then for 3 more doses every 6 hours.
  Epidural Morphine: All patients, including those in both the experimental and control groups, in this study will receive epidural morphine prior to removal of epidural catheter as part of routine obstetric care for cesarean delivery.
  Hydromorphone: Post-operatively all patients patients will have intravenous hydromorphone on an as needed basis to control their pain, as part of routine obstetric care for cesarean delivery.
Period: Overall Study
Arm/Group | Ketorolac | Placebo
Started | 35 | 35
Intraoperative Checkpoint (Checkpoint to confirm patients still meet inclusion and exclusion criteria.) | 28 | 30
Completed | 28 | 30
Not Completed | 7 | 5
Not completed — Cesarean after 4pm / Unable to complete enrollment due to floor acuity | 5 | 3
Not completed — Obstetrician refusal | 0 | 1
Not completed — Patient elected for TOLAC | 1 | 0
Not completed — Cesarean deemed stat | 1 | 0
Not completed — Anaphylaxis prior to cord clamp to non-study drug | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketorolac | Placebo | Total
Number analyzed (Participants) | 28 | 30 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (5.4) | 27.4 (5.5) | 28.1 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 30 | 58
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 17 | 36
  White | 8 | 10 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Weight (kg) [Mean (Standard Deviation); unit: kg] | 100.0 (24.7) | 93.8 (25.1) | 96.8 (24.9)
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m^2] | 38.1 (8.5) | 35.1 (8.2) | 36.5 (8.4)
Gravida [Median (Inter-Quartile Range); unit: prior pregnancies] | 3 [2 to 3] | 2.5 [2 to 3] | 3 [2 to 3]
Parity [Mean (Standard Deviation); unit: births carried to viability] | 1.3 (0.8) | 1.1 (0.8) | 1.2 (0.8)
Prior Cesarean delivery (CD) [Median (Inter-Quartile Range); unit: prior Cesareans] | 1 [1 to 1.5] | 1 [0 to 2] | 1 [1 to 2]
Tubal Ligation at time of CD [Count of Participants; unit: Participants] | 12 | 6 | 18
Preoperative Hematocrit (Hct) [Mean (Standard Deviation); unit: mg/dl] | 34.6 (3.0) | 34.2 (3.0) | 34.4 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Estimated Blood Loss (EBL)
Description: Estimation of blood loss during surgery
Time Frame: Immediately post-op
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Ketorolac | Placebo
Number analyzed (Participants) | 28 | 30
ml | 900 [692.5 to 1047] | 800 [600 to 1000]
Statistical Analysis 1: Comparison: Ketorolac vs Placebo; Test type: Superiority; p = 0.34, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Post-Partum Hemorrhage
Description: Rate of Post-Partum Hemorrhage between groups during the first 24 hours pst-partum.
Time Frame: 0 - 24 hours post-partum
Measure: Count of Participants; unit: Participants
Groups:
- Ketorolac: Patients in this arm will be given ketorolac at cord clamp with standard dose of 30 mg, then 3 additional 30 mg doses every 6 hours
  Ketorolac: Patients in the experimental arm will receive ketorolac 30 mg in 1 ml at the time of cord clamp and then for 3 more doses every 6 hours.
- Placebo: Patients in this arm will be given a placebo medication at cord clamp, and then 3 additional doses of placebo every 6 hours.
  Normal Saline: Patients in the control arm will receive normal saline 1 ml at the time of cord clamp and then for 3 more doses every 6 hours.
Arm/Group | Ketorolac | Placebo
Number analyzed (Participants) | 28 | 30
Participants | 7 | 4
Statistical Analysis 1: Comparison: Ketorolac vs Placebo; Test type: Superiority; p = .257, Chi-squared

3. Secondary Outcome: Corrected Change in Hct on POD1.
Description: Corrected change in Hct on POD1. Performed by subtracting POD1 Hct from POD0 Hct. Correction for transfusion by further subtracting 3 per unit of pRBC transfused to account for the typical change seen per unit transfused.
Time Frame: POD1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Ketorolac | Placebo
Number analyzed (Participants) | 28 | 30
mg/dl | -5.1 (3.5) | -3.5 (3.6)
Statistical Analysis 1: Comparison: Ketorolac vs Placebo; Test type: Superiority; p = 0.085, t-test, 2 sided

4. Secondary Outcome: Uterotonic Doses
Description: Total number of uterotonic doses including methylergonovine, carboprost and misoprostol.
Time Frame: 0 - 24 hours post-partum
Measure: Median (Inter-Quartile Range); unit: doses
Arm/Group | Ketorolac | Placebo
Number analyzed (Participants) | 28 | 30
doses | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Ketorolac vs Placebo; Test type: Superiority; p = 0.164, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Units of Packed Reb Blood Cell Transfused
Description: Total number of Units of Packed Reb Blood Cell Transfused in intra-op until 24 hours post-partum.
Time Frame: Intra-op until 24 hours post-partum.
Measure: Median (Inter-Quartile Range); unit: units of pRBCs
Arm/Group | Ketorolac | Placebo
Number analyzed (Participants) | 28 | 30
units of pRBCs | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Ketorolac vs Placebo; Test type: Superiority; p = 1.000, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Hydromorphone Use
Description: Use of any intravenous hydromorphone administered within the first 24 hours after cesarean delivery.
Time Frame: 0 - 24 hours post-partum
Measure: Count of Participants; unit: Participants
Arm/Group | Ketorolac | Placebo
Number analyzed (Participants) | 28 | 30
Participants
  Non-use of Opioids | 17 | 10
  Use of Opioids | 11 | 20
Statistical Analysis 1: Comparison: Ketorolac vs Placebo; Test type: Superiority; p = 0.0367, Chi-squared; Risk Difference (RD) = -0.27, 95% CI 2-sided [-0.52 to -0.03]

7. Secondary Outcome: Total Hydromorphone Dose
Description: Total hydromorphone doses in mg in the first 24 hours post-partum.
Time Frame: 0 - 24 hours post-partum.
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Ketorolac | Placebo
Number analyzed (Participants) | 28 | 30
mg | 0 [0 to 0.2] | 0.2 [0 to 0.4]
Statistical Analysis 1: Comparison: Ketorolac vs Placebo; Test type: Superiority; p = 0.0231, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Anti-emetic Doses
Description: Total doses of medications to treat pruritus (opioid side-effect) including ondansetron and promethazine.
Time Frame: 0 - 24 hours post-partum
Measure: Median (Inter-Quartile Range); unit: doses
Arm/Group | Ketorolac | Placebo
Number analyzed (Participants) | 28 | 30
doses | 0 [0 to 1] | 0 [0 to 1]
Statistical Analysis 1: Comparison: Ketorolac vs Placebo; Test type: Superiority; p = 0.467, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Pruritus Doses
Description: Total doses of medications to treat pruritus (opioid side-effect) including diphenhydramine, nalbuphine and naloxone.
Time Frame: 0 - 24 hours post-partum
Measure: Median (Inter-Quartile Range); unit: doses
Arm/Group | Ketorolac | Placebo
Number analyzed (Participants) | 28 | 30
doses | 0 [0 to 1] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Ketorolac vs Placebo; Test type: Superiority; p = 0.273, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Percentile Change in Systolic Blood Pressure at 6,12, and 24 Hours
Description: Percentile change in Systolic Blood Pressure at 6,12, and 24 hours for each patient's baseline defined by immediate post-op PACU vitals.
Time Frame: 0 - 24 hours post-partum
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ketorolac | Placebo
Number analyzed (Participants) | 28 | 30
Percent change
  6 hours | -2.0 (11.6) | -0.6 (10.00)
  12 hours | -9.10 (8.99) | -2.85 (10.13)
  24 hours | -5.9 (12.4) | -3.5 (12.2)
Statistical Analysis 1: Comparison: Ketorolac vs Placebo; Test type: Superiority; p = 0.0162, t-test, 2 sided — p-value for 12 hours post-op between-group comparison

11. Secondary Outcome: Percentile Change in Diastolic Blood Pressure (DBP) at 6,12, and 24 Hours
Description: Percentile change in diastolic Blood Pressure at 6,12, and 24 hours for each patient's baseline defined by immediate post-op PACU vitals.
Time Frame: 0 - 24 hours post-partum
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ketorolac | Placebo
Number analyzed (Participants) | 28 | 30
Percent change
  6 hours | 12.30 (17.7) | 7.6 (17.6)
  12 hours | 8.8 (17.3) | 8.8 (16.2)
  24 hours | 12.0 (19.4) | 11.1 (22.2)

12. Secondary Outcome: Change in Pain Score Post-Cesarean Delivery
Description: Pain score post-Cesarean Delivery using 11-point numerical rating scale (NRS): 0-10 where 0 is no pain and 10 is the worst pain imaginable
Time Frame: Up to 24 hours post-cesarean delivery
Measure: Median (Inter-Quartile Range); unit: units on NRS
Arm/Group | Ketorolac | Placebo
Number analyzed (Participants) | 28 | 30
units on NRS
  Baseline | 0 [0 to 0] | 0 [0 to 0]
  15 mins | 0 [0 to 0] | 0 [0 to 0]
  1 hour | 0 [0 to 3] | 0 [0 to 6]
  6 hours | 1 [0 to 4.5] | 3 [1 to 6]
  12 hours | 2 [0 to 4.5] | 3.5 [1 to 5]
  24 hours | 4.5 [2.5 to 6.5] | 5.5 [3 to 7]
Statistical Analysis 1: Comparison: Ketorolac vs Placebo; Test type: Superiority; p = 0.048, Wilcoxon (Mann-Whitney) — p-value for 6 hours post-op between-group comparison

ADVERSE EVENTS:
Time Frame: Patients were followed throughout their hospital stay to monitor for any adverse events. Post cesarean delivery hospital stay is typically 3-4 days. No monitoring for adverse events occurred after discharge.
Arm/Group | Ketorolac | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/30
Other Adverse Events (participants affected / at risk) | 0/28 | 0/30

LIMITATIONS AND CAVEATS:
Limitations include:

* single-center study.
* secondary outcomes may not fully represent opioid-sparing and pain seen in a center practicing current SOAP ERAC protocol as patients received epidural and not intrathecal morphine and not all patients received all doses of acetaminophen.
* secondary outcomes may not fully represent the opioid-sparing and pain effects of ketorolac, as not all ketorolac patients received all doses of ketorolac.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-28): https://cdn.clinicaltrials.gov/large-docs/12/NCT02509312/Prot_SAP_000.pdf